CLINICAL TRIAL: NCT02435823
Title: Adjunctive Wide-neck Aneurysm Reconstruction Device Post Market Clinical Study Europe
Brief Title: Safety Study of the PulseRider® in Patients Undergoing Treatment for Bifurcation Intracranial Aneurysms
Acronym: AWARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulsar Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0015
Record Dates: First submitted 2015-04-28; First posted 2015-05-06 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Brain Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PulseRider (Experimental): Endovascular treatment of intracranial aneurysms
  Interventions: Device: PulseRider

INTERVENTIONS:
Device: PulseRider — Adjunctive device for endovascular embolization of intracranial aneurysms

SUMMARY:
This is a prospective multi-center, single arm, non-randomized study. It is designed to evaluate the safety of the PulseRider® in patients undergoing treatment for bifurcation intracranial aneurysms.

DETAILED DESCRIPTION:
Primary Endpoints:

Safety: Death or stroke in downstream territory to 180-days post-procedure Technical Success: Device placement success and ability to retain coils within the aneurysm (as judged by the treating physician at the time of the procedure. Core lab will review images at a later time) Rate of aneurysm occlusion at Day zero (0) and 180-days

Additional Evaluations to 180-days and at 365-day follow up Rate of aneurysm occlusion at 365 days Device movement or migration defined as any relative change in the position of the device with respect to the parent and/or daughter vessels that is greater than 2mm by conventional catheter angiography, CTA or MRA (180 days) and (365 days) Stenosis defined as >50% at implant site by conventional catheter angiography, MRA or CTA at 180 days and at 365 days Rate of incidence of new neurological deficits Complication rate (neurological and non-neurological)

ELIGIBILITY:
Inclusion Criteria:

1. Patient who presents with an MRA, CTA or angiographically confirmed, wide neck (> 4 mm or dome to neck ratio < 2) intracranial aneurysms located at a bifurcation
2. The target aneurysm is in a vessel with a diameter of 2.7 mm to 4.5mm.
3. The patient is 18 years or older at the time of consent
4. The patient has signed the IRB/EC approved informed consent form
5. In the opinion of the physician, placement of the PulseRider is technically feasible and clinically indicated
6. Subject has mental capacity and is willing and able to comply with protocol requirements and follow-up

Exclusion Criteria:

1. Unstable neurological deficit (condition worsening within the last 90 days)
2. Subarachnoid Hemorrhage (SAH) within the last 60 days
3. Irreversible bleeding disorder
4. mRS score ≥3
5. Patient has another aneurysm which, in the Investigator's opinion, will require treatment within the follow up period (365 days)
6. Platelet count < 100 x 103 cells/mm3or known platelet dysfunction
7. Inability to tolerate, adverse reaction or contraindication to taking aspirin or clopidogrel
8. A history of contrast allergy that cannot be medically controlled
9. Known allergy to nickel
10. Relative contraindication to angiography (e.g., serum creatinine > 2.5 mg/dL)
11. Woman with child-bearing potential who cannot provide a negative pregnancy test
12. Evidence of active infection (fever with temperature > 38°C and/or WBC > 15,000)
13. Other conditions of the heart, blood, brain or intracranial vessels that carry a high risk of neurologic events
14. Evidence of disease or condition expected to compromise survival or ability to complete follow-up assessments during the 365-day follow-up period
15. Extracranial stenosis greater than 50% in the parent artery requiring access to the lesion
16. Intracranial stenosis greater than 50% in the treated vessel
17. Extreme vessel tortuosity that prohibits appropriate control of the micro-guide wire and/or the PulseRider delivery wire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2015-03-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Safety: Death or stroke in downstream territory | to 180-days post-procedure
Technical Success | at the time of the procedure
  Device placement success and ability to retain coils within the aneurysm
Rate of aneurysm occlusion | Day zero (within 24 hours post procedure) and 180-days

SECONDARY OUTCOMES:
Rate of aneurysm occlusion | at 365-days follow-up
Device movement or migration defined as any relative change in the position of the device with respect to the parent and/or daughter vessels that is greater than 2mm by conventional catheter angiography, MRA or CTA | at 180-days follow-up and 365-days follow-up
Stenosis, defined as >50% at implant site by MR angiography or conventional catheter angiography or CTA | at 180-days follow-up and 365-days follow-up
Rate of incidence of new neurological deficits | from the time of the procedure to the 365-follow up visit
Complication rate (neurological and non-neurological) | from the time of the procedure to the 365-follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Monika Killer, MD, Principal Investigator — Paracelsus Medical University
Locations (1):
- Paracelsus Medical University Salzburg, Salzburg, Austria